CLINICAL TRIAL: NCT02573740
Title: A Study to Evaluate the Safety, Tolerability and the Effects on Cerebrospinal Fluid Spectrin Breakdown Product-145 Levels of Multiple Doses of ABT-957 in Subjects With Mild Alzheimer's Disease and Mild Cognitive Impairment Due to Alzheimer's Disease
Brief Title: Safety, Tolerability and the Effects on Cerebrospinal Fluid Spectrin Breakdown Product-145 Levels of ABT-957 in Subjects With Mild Alzheimer's Disease and Mild Cognitive Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient target engagement of ABT-957 (preclinical data)
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M13-730
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — alicapistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-957 (Experimental): ABT-957 given twice a day for 84 days
  Interventions: Drug: ABT-957
- Placebo (Placebo Comparator): Placebo given twice a day for 84 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ABT-957
  Arms: ABT-957
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1, multicenter, randomized, double-blind, placebo-controlled, multiple dose study of ABT-957 in participants with mild Alzheimer's disease (AD) and Mild Cognitive Impairment (MCI) due to AD.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must have negative results for pregnancy test performed on a serum sample obtained at Screening
* Body Mass Index is 18.0 to 35.0 at Screening
* Meets the National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria for probable Alzheimer's disease (AD).
* Meets the NIA-AA core clinical criteria for Mild Cognitive Impairment due to AD

Exclusion Criteria:

* Use of any strong inhibitors of drug metabolizing enzymes within 30 days prior to study drug administration
* Consumption of alcohol within 24 hours prior to study drug administration
* Positive screen for non-prescribed drugs of abuse or alcohol
* The participant has clinically significant abnormal laboratory values at Screening as determined by the investigator
* History of a drug or alcohol abuse within 6 months prior to study drug administration
* Current diagnosis of major depression or other major psychiatric disorder

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting treatment-emergent adverse events | For approximately 84 days
Level of spectrin breakdown product-145 (SBDP-145) | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Nuno Mendonca, MD, Study Director — AbbVie
Locations (9):
- United States (9):
  - Site Reference ID/Investigator# 143180, Cypress, California
  - Site Reference ID/Investigator# 143178, Orlando, Florida
  - Site Reference ID/Investigator# 149484, The Villages, Florida
  - Site Reference ID/Investigator# 143181, Marlton, New Jersey
  - Site Reference ID/Investigator# 143182, Cincinnati, Ohio
  - Site Reference ID/Investigator# 149481, Dallas, Texas
  - Site Reference ID/Investigator# 143254, Orem, Utah
  - Site Reference ID/Investigator# 143179, Salt Lake City, Utah
  - Site Reference ID/Investigator# 143177, Spokane, Washington

REFERENCES:
- [Result] Lon HK, Mendonca N, Goss S, Othman AA, Locke C, Jin Z, Rendenbach-Mueller B. Pharmacokinetics, Safety, Tolerability, and Pharmacodynamics of Alicapistat, a Selective Inhibitor of Human Calpains 1 and 2 for the Treatment of Alzheimer Disease: An Overview of Phase 1 Studies. Clin Pharmacol Drug Dev. 2019 Apr;8(3):290-303. doi: 10.1002/cpdd.598. Epub 2018 Jul 27. PMID 30052328